CLINICAL TRIAL: NCT05960760
Title: Assessing the Cross-cultural Validity and Reliability of the German Version of the Back Pain Attitudes Questionnaire (Back-PAQ_G) Within the German-speaking Swiss Population
Brief Title: Attitudes Towards Back and Back Pain in German-speaking Switzerland
Status: Completed | Type: Observational
Sponsor: Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Fabian Pfeiffer, PT, MSc, Zurich University of Applied Sciences
Other Study IDs: Back-PAQ_G
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research aims to assess the cross-cultural validity and reliability of the German version of the Back-PAQ (Back-PAQ_G) within the German-speaking Swiss population.

The target population for this study includes individuals with and without back pain and primary care healthcare professionals. This includes physicians, physiotherapists, and nurses. The participants will be asked to fill out the Back-PAQ_G and similiar questionnaires online.

ELIGIBILITY:
Inclusion Criteria:

* Living within the German-speaking part of Switzerland

Exclusion Criteria:

* Insufficient German language skills

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population for this study includes individuals with and without back pain and primary care healthcare professionals. This includes physicians, physiotherapists, and nurses.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Back Pain and Attitudes Questionnaire | baseline
  The Back-PAQ_G contains 34 statements about the lower back and back pain that have to be rated as "true", "uncertain" or "false". Scores range from 34 to 170. The higher the score, the more unhelpful attitudes toward the back and back pain are present. Participants will receive the German version of the Back-PAQ (Back-PAQ_G).

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia | baseline
  The TSK examines fear of movement and injury. The TSK applies to individuals with and without pain. The scores range from 11 to 44. A higher score on the completed questionnaire implies high kinesiophobia and an existing somatic focus. The participants of the study receive the German version of TSK-GV with eleven questions.
Fear Avoidance Belief Questionnaire | baseline
  The FABQ examines fear avoidance attitudes about the effect of work and activity on lower back pain. The questionnaire applies to individuals with low back pain. The maximum score is 96. A high score indicates a strong fear-avoidance posture for low back pain. Participants with current low back pain receive the validated German version of the FABQ with 16 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Pfeiffer, MSc, Principal Investigator — ZHAW, Department Gesundheit, Institut für Physiotherapie
Locations (2):
- Switzerland (2):
  - 4 Balance Zentrum für Physiotherapie und medizinisches Training, Muttenz, Basel-Landschaft
  - Kantonsspital Winterthur (KSW), Winterthur

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Darlow B, Perry M, Mathieson F, Stanley J, Melloh M, Marsh R, Baxter GD, Dowell A. The development and exploratory analysis of the Back Pain Attitudes Questionnaire (Back-PAQ). BMJ Open. 2014 May 23;4(5):e005251. doi: 10.1136/bmjopen-2014-005251. PMID 24860003